CLINICAL TRIAL: NCT01345578
Title: Hepatocyte Transplantation for Liver Based Metabolic Disorders
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: seeking additional funding
Sponsor: Ira Fox (Other)
Responsible Party: Sponsor-Investigator, Ira Fox, Professor of Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO09040497
Record Dates: First submitted 2011-04-26; First posted 2011-05-02 (Estimated); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Metabolic Diseases
Keywords: Urea Cycle Disorders; Carbamoyl-Phosphate Synthase I Deficiency Disease; Citrullinemia; Ornithine Carbamoyltransferase Deficiency Disease; Crigler-Najjar Syndrome
MeSH Terms: conditions — Metabolic Diseases; Urea Cycle Disorders, Inborn; Carbamoyl-Phosphate Synthase I Deficiency Disease; Citrullinemia; Ornithine Carbamoyltransferase Deficiency Disease; Crigler-Najjar Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hepatocyte Transplantation (Experimental): See Below
  Interventions: Drug: human hepatocyte transplantation; Radiation: Preparative Radiation Therapy

INTERVENTIONS:
Drug: human hepatocyte transplantation — Transplantation of hepatocytes into the liver will be through the portal vein. The portal vein will be accessed transhepatically, by umbilical vein, or surgically by a peripheral mesenteric vein.
  The subject will be evaluated de novo and if they are a candidate for orthotopic liver transplantation they will receive the transplant. Even if the subject receives the hepatocyte transplant and it does not work, they will be evaluated for orthotopic liver transplantation as if they never received the hepatocyte transplant.
  If at 6 months we see an improvement in disease, we will recommend a re-transplantation with a goal of complete correction of disease and until the subject is no longer required to be a candidate for organ transplantation. Subjects will be re-evaluated every 6 months for re-transplantation. Subjects will remain on the waiting list for organ transplantation. Further radiation therapy will not be needed prior to re-transplantation.
  Other Names: hepatocyte transplant
Radiation: Preparative Radiation Therapy — Just prior to the hepatocyte transplant, a portion of the right hepatic lobe comprising between 35-50% of the entire liver volume will be irradiated to a dose of 7.5-10 Gy in a single fraction using a linear accelerator-based stereotactic radiosurgery system with intensity-modulated radiation therapy planning (IMRT).

SUMMARY:
The purpose of this research study is to determine whether partial irradiation of the liver and liver cell transplantation can provide help for patients with life-threatening liver-based metabolic diseases who are unlikely to survive without extensive medical therapy or transplant. The goal of this research study is to determine if liver cell transplants can be effective as an alternative to organ transplantation. At the present time, liver cell transplants are experimental and have been done in a limited number of human subjects.

DETAILED DESCRIPTION:
Management of patients with hepatic failure and liver-based metabolic disorders is complex and expensive. Hepatic failure results in impaired coagulation, altered consciousness and cerebral function, a heightened risk of multiple organ system failure, and sepsis. Liver transplantation is often the only available treatment option for severe, even if transient, hepatic failure. Patients with life-threatening liver-based metabolic disorders similarly require organ transplantation even though their metabolic diseases are typically the result of a single enzyme deficiency, and the liver otherwise functions normally. More than 17,000 patients currently await liver transplantation in the United States, a number that seriously underestimates the number of patients that need treatment, as it has been estimated that more than a million patients in the United States could benefit from transplantation. Unfortunately, use of whole liver transplantation to treat these disorders is limited by a severe shortage of donors and by the risks associated with major surgery. Hepatocyte transplantation holds great promise as an alternative to organ transplantation for the treatment of liver diseases, and numerous studies in rodents indicate that transplants consisting of isolated liver cells can correct various metabolic deficiencies of the liver and can reverse hepatic failure. The transplant procedure, which involves injection of isolated hepatocytes into the liver through the portal vein, is far less intrusive than transplantation of the whole liver and could be performed on severely ill patients with relatively low risk. In the presence of normal host liver architecture, the transplanted cells integrate into the host liver, providing considerable restorative potential. Because the native liver is not removed, the transplanted hepatocytes need only improve some of the functions of the failing liver and need not replace all hepatic functions. Although clinical trials of hepatocyte transplantation have demonstrated the long-term safety of the procedure, only partial correction of metabolic disorders has been achieved, and the degree to which donor hepatocytes have restored failing livers has not been adequate to circumvent the need for organ replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have life-threatening liver-based metabolic disorders who are candidates for organ transplantation where hepatocyte transplantation is considered theoretically curative.
* In addition to child subjects less than 18 years of age, for purposes of this protocol, adults up to age 21 years will be enrolled since this is the upper age limit of patients which are seen at Children's Hospital of Pittsburgh.

Exclusion Criteria:

* Patients with liver based metabolic disorders not theoretically treatable with organ transplantation.
* Subjects who meet any of the following criteria will be excluded from participation in this protocol:

  1. Subject has active malignancy.
  2. Subject has allergy to immunosuppression medications that are required post transplant procedure for the prevention of rejection.
  3. Subject has sepsis, pneumonia, other active infection or other secondary life-threatening organ dysfunction.
  4. Significant liver fibrosis determined by biopsy (if clinically indicated). Significant liver fibrosis will be defined by the Ishak Staging, Stage 5: bridges with occasional nodules.
  5. Subject is pregnant or breastfeeding.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2011-03; Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Improvement in enzyme physiologic function at 6 months | 6 months post hepatocyte transplant
  After infusing donor allogeneic hepatocytes through the portal vein following preparative hepatic irradiation, improvement in enzyme physiologic function will be assessed at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ira J Fox, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Horslen SP, Fox IJ. Hepatocyte transplantation. Transplantation. 2004 May 27;77(10):1481-6. doi: 10.1097/01.tp.0000113809.53415.c2. PMID 15239608
- [Background] Horslen SP, McCowan TC, Goertzen TC, Warkentin PI, Cai HB, Strom SC, Fox IJ. Isolated hepatocyte transplantation in an infant with a severe urea cycle disorder. Pediatrics. 2003 Jun;111(6 Pt 1):1262-7. doi: 10.1542/peds.111.6.1262. PMID 12777539
- [Background] Fox IJ, Chowdhury JR, Kaufman SS, Goertzen TC, Chowdhury NR, Warkentin PI, Dorko K, Sauter BV, Strom SC. Treatment of the Crigler-Najjar syndrome type I with hepatocyte transplantation. N Engl J Med. 1998 May 14;338(20):1422-6. doi: 10.1056/NEJM199805143382004. No abstract available. PMID 9580649
- [Background] Dhawan A, Mitry RR, Hughes RD, Lehec S, Terry C, Bansal S, Arya R, Wade JJ, Verma A, Heaton ND, Rela M, Mieli-Vergani G. Hepatocyte transplantation for inherited factor VII deficiency. Transplantation. 2004 Dec 27;78(12):1812-4. doi: 10.1097/01.tp.0000146386.77076.47. PMID 15614156
- [Background] Sokal EM, Smets F, Bourgois A, Van Maldergem L, Buts JP, Reding R, Bernard Otte J, Evrard V, Latinne D, Vincent MF, Moser A, Soriano HE. Hepatocyte transplantation in a 4-year-old girl with peroxisomal biogenesis disease: technique, safety, and metabolic follow-up. Transplantation. 2003 Aug 27;76(4):735-8. doi: 10.1097/01.TP.0000077420.81365.53. PMID 12973120
- [Derived] Jorns C, Ellis EC, Nowak G, Fischler B, Nemeth A, Strom SC, Ericzon BG. Hepatocyte transplantation for inherited metabolic diseases of the liver. J Intern Med. 2012 Sep;272(3):201-23. doi: 10.1111/j.1365-2796.2012.02574.x. Epub 2012 Aug 20. PMID 22789058